CLINICAL TRIAL: NCT00457665
Title: Mecahnisms of Lipodystrophy in HIV-Infected Patients
Brief Title: Mechanisms of Lipodystrophy in HIV-Infected Pateints
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01-56583
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-05

CONDITIONS: HIV Infections
Keywords: HIV; Lipodystrophy; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — Nelfinavir; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nelfinavir (Viracept) (Active Comparator)
  Interventions: Drug: Nelfinavir
- Efavirenz (Sustiva) (Active Comparator)
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Nelfinavir
  Other Names: Viracept
  Arms: Nelfinavir (Viracept)
Drug: Efavirenz
  Arms: Efavirenz (Sustiva)

SUMMARY:
The metabolic and molecular basis of lipodystrophy syndrome in HIV-infected patients is not known. Whether besides protease inhibitors, other antiretroviral drugs, HIV infection and reduction in viral load contribute to the development of lipodystrophy syndrome is not clear.

The project therefore has the following aims: 1) to characterize metabolic abnormalities and changes in body fat distribution, 2) to develop objective criteria for defining the syndrome and to ascertain prognostic indicators and 3) to elucidate the molecular basis of the lipodystrophy syndrome in HIV-infected patients.

DETAILED DESCRIPTION:
A 2-year long prospective, randomized, double blind, placebo-controlled study in 200 asymptomatic HIV (+) patients to compare two equally effective antiretroviral regimens, one with and the other without a protease inhibiotor. We will study body fat distribution by anthropometry and magnetic resonance imaging and will measure insulin sensitivity (in a subset of patients), plasma lipoproteins, glucose tolerance and other metabolic variables. We will study expression of an array of adipocyte specific proteins/transcription factors involved in adipocyte differentiation, insulin action and lipoprotein metabolism in fat biopsy samples obtained before and after institution of therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV Positive
* No previous antiviral therapy
* 18 to 70 years of age

Exclusion Criteria:

* Patients with opportunistic infections or AIDS.
* Active intravenous drug users.
* Patients on corticosteroids, androgens, lipid-lowering drugs, anti-fungal medications, dehydroepiandrosterone, oxandrolone, megace.
* Patients with diabetes mellitus.
* Patients with moderate to heavy alcohol consumption ( greater than 15 drinks per week).
* Pregnant or premenopausal women, unless surgically sterilized or highly unlikely to conceive (defined as women taking oral contraceptives, using barrier protection during intercourse or with a copper intrauterine device in place for > 3 months without complaints and a negative serum or urine pregnancy test within 30 days of study entry).
* Acute or chronic liver diseases; elevations of liver transaminases by more than two and one half times above the upper limits of normal ( SGOT > 105 U/L, SGPT > 120 U/L, ) or a total bilirubin of > 1.5mg/dL.
* Anemia (hematocrit <32%).
* Abnormal thyroid function tests.
* Weight loss >10% from baseline in the past year.
* Recent (within the past year), history of suicide attempt.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-02; Primary Completion 2007-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, M.D., Principal Investigator — University of Texas Southwestern Medical Center Dallas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nelfinavir: Randomized to receive Nelfinavir inclusive HAART
- Efavirenz: Randomized to receive Efavirenz inclusive HAART
Period: 12 Months
Arm/Group | Nelfinavir | Efavirenz
Started | 28 | 28
Completed | 20 | 19
Not Completed | 8 | 9
Not completed — Drug allergy | 1 | 1
Not completed — High HIV viral load | 5 | 1
Not completed — Lipodystrophy | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Abnormal Liver function tests | 0 | 5
Period: 24 Months
Arm/Group | Nelfinavir | Efavirenz
Started | 20 | 19
Completed | 15 | 11
Not Completed | 5 | 8
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lipodystrophy | 1 | 1
Not completed — Abnormal liver function tests | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nelfinavir | Efavirenz | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 23 | 24 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 14 | 19 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 13
Weight [Mean (Standard Deviation); unit: kgs] | 75.4 (11) | 75 (13.8) | 75.18 (12.3)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.2 (3.8) | 24.8 (5) | 24.9 (4.3)
CD4 count [Mean (Standard Deviation); unit: per cubic mm] — Population: Data for 2 patients were not available
  per cubic mm
    number analyzed (Participants) | 28 | 26 | 54
    (all) | 312 (210) | 301 (158) | 307 (185)
HIV Viral load [Median (Full Range); unit: copies per mL] — Population: Values for 3 participants were not available
  copies per mL
    number analyzed (Participants) | 28 | 25 | 53
    (all) | 82000 [6230 to 750001] | 103000 [5220 to 750001] | 97900 [5220 to 750001]
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] — Population: Values of 3 participants were not available
  mg/dL
    number analyzed (Participants) | 26 | 27 | 53
    (all) | 92.5 (9.0) | 90.3 (5.6) | 91.4 (7.4)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 129 (83.8) | 133.5 (81.4) | 131.24 (82)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Drug Regimens on Serum Triglycerides.
Time Frame: 12 and 24 months
Population: Some subjects dropped before 1 year and some dropped between 1-2 years.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Nelfinavir (Viracept): Assigned to Nelfinavir
- Efavirenz (Sustiva): Assigned to Efavirenz
Arm/Group | Nelfinavir (Viracept) | Efavirenz (Sustiva)
Number analyzed (Participants) | 20 | 20
mg/dL
  At 12 months | 228.0 (119.0) | 230.4 (157.3)
  At 24 months: number analyzed (Participants) | 14 | 11
  At 24 months | 293.4 (350.6) | 290.0 (276.1)
Statistical Analysis 1: Comparison: Nelfinavir (Viracept) vs Efavirenz (Sustiva); Test type: Superiority; p = 0.94, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Nelfinavir: These participants were randomized to receive Nelfinavir
- Efavirenz: These participants were randomized to receive Efavirenz
Arm/Group | Nelfinavir | Efavirenz
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 2/28
Other Adverse Events (participants affected / at risk) | 20/28 | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfinavir (N=28) | Efavirenz (N=28)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalized
Vomiting and diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalized
Spider bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Hospitalized
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfinavir (N=28) | Efavirenz (N=28)
Peripheral neuropathy (Nervous system disorders) | 6 (6) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 13 | 1
Abnormal liver function tests (Hepatobiliary disorders) | 1 (1) | 10 (10) — High values of aspartate aminotransferase or alanine aminotransferase
Disturbing dreams (Psychiatric disorders) | 2 | 9
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes